CLINICAL TRIAL: NCT03319420
Title: A Randomized, Double-Masked, Comparative Study Versus Systane Ultra UD, to Evaluate the Efficacy and Safety of LO2A Eye Drops for Symptomatic Improvement of Dry Eye in Patients With Sjögren's Syndrome
Brief Title: Evaluate the Efficacy and Safety of LO2A Eye Drops for Symptomatic Improvement of Dry Eye in Patients With Sjögren's Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ocuwize LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WP-LO2A-03
Record Dates: First submitted 2017-10-19; First posted 2017-10-24 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2019-07

CONDITIONS: Dry Eye Due to Sjögren's Syndrome

STUDY DESIGN:
Intervention Model Description: A randomized, double-Masked, comparative study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Investigator staff involved in the dispensation of study treatments and treatment compliance checks will not be involved in data collection - doublemasked treatment design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LO2A (Experimental): 1 drop of sodium hyaluronate instilled into each eye 4 times daily
  Interventions: Drug: LO2A eye drops
- Systane Ultra UD (Active Comparator): 1 drop of Systane Ultra UD instilled into each eye 4 times daily
  Interventions: Drug: Systane Ultra UD

INTERVENTIONS:
Drug: LO2A eye drops — Sodium hyaluronate
  Arms: LO2A
Drug: Systane Ultra UD — Active Ingredients; Polyethylene Glycol Propylene Glycol
  Arms: Systane Ultra UD

SUMMARY:
Dry eye complaints occur in 5.5 to 33.7% of the population, and are ranked as the most frequent symptoms of patients visiting ophthalmologists. Dry eye syndrome is caused by the reduced production and/or improper quality of the tear film. One of the causes of reduced tear production is Sjögren's syndrome. Sjögren's is estimated to affect up to 4 million patients in the US alone. It affects mostly middle aged women (40-50 years of age) with a female to male prevalence ratio of 9:1.

The current study seeks to evaluate the safety and efficacy of LO2A ophthalmic solution in the symptomatic treatment of dry eye in patients with Sjögren's syndrome. This study will be conducted in compliance with the protocol, GCP,and applicable regulatory requirements.

DETAILED DESCRIPTION:
This is a randomized, double-masked, comparative study versus Systane ultra UD, to evaluate the efficacy and safety of LO2A eye drops for symptomatic improvement of dry eye in Patients with Sjögren's syndrome. Eligible patients will be randomly assigned in a 1:1 ratio to one of two treatment groups, LO2A or Systane ultra UD, respectively.

The study will consist of a screening period of up to two weeks and a 3-month double blind treatment period (topical application of eye drops four times daily)

Up to 60 subjects are planned to be recruited to this study, randomized to one of two treatment arms using a 1:1 active (LO2A) to Systane ultra UD ratio.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any race and ≥ 18 years of age.
* Willing and able to provide voluntary written informed consent.
* Primary or secondary Sjögren's syndrome according to the American- European Consensus Classification Criteria (2002).
* Females of childbearing potential must agree to use effective contraception consistently throughout the study (such as hormonal contraception or two forms of barrier contraception) and have a negative urine pregnancy test at screening.
* Willing and able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* Subject has concurrent, uncontrolled medical condition, or psychiatric illness which could place him/her at unacceptable risk.
* Subjects with pterygium.
* Subjects with active, allergic keratoconjunctivitis, or conjunctivitis of infectious origin.
* Subjects with blepharitis requiring treatment.
* Subjects with a history of surgery affecting the eye surface, as well as eye injuries within 3 months of screening.
* Subjects currently using any topical ophthalmic treatment (including medications for glaucoma) or over-the-counter (OTC) solutions, artificial tears, gels or scrubs, and cannot discontinue these medications for the duration of the trial.
* Female subjects who are pregnant or breast-feeding, or plan to become pregnant during the study.
* Subjects that have started or changed the dose of chronic systemic medication within 7 days of Visit 1.
* Known hypersensitivity to sodium hyaluronate or any LO2A excipients (glycerol and Carbomer 981) or any of the components in Systane Ultra UD.
* Active abuse of alcohol or drugs.
* Any condition, which in the opinion of the Investigator, would place the patient at an unacceptable risk if participating in the study protocol.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2021-01-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Change in corneal / conjunctival staining score using the National Eye Institute/Industry(NEI) Industry Grading System | 3 months form the basline
  NEI/Industry Workshop Conjunctival Staining Grading System. Devitalized epithelial cells of the bulbar conjunctiva are stained with lissamine green and can graded across six zones The scores for each zone (0-3) are summed to obtain an overall score for each eye (0-18.( The higher the results, the more severe the dryness of the eye.

SECONDARY OUTCOMES:
Change in Ocular Surface Disease Index (OSDI) questionnaire score. | 1 and 3 months from the basline visit
  The OSDI is assessed on a scale of 0 to 100, with higher scores representing greater disability. The index demonstrates sensitivity and specificity in distinguishing between normal subjects and patients with dry eye disease.
Change in corneal / conjunctival staining score using the National Eye Institute/Industry(NEI) Industry Grading System | After one month
  NEI/Industry Workshop Conjunctival Staining Grading System. Devitalized epithelial cells of the bulbar conjunctiva are stained with lissamine green and can graded across six zones The scores for each zone (0-3) are summed to obtain an overall score for each eye (0-18.( The higher the results, the more severe the dryness of the eye.

CONTACTS AND LOCATIONS:
Locations (5):
- Israel (5):
  - HaEmek MC, Afula
  - Rambam, Haifa
  - Rabin MC, Petah Tikva
  - Kaplan MC, Rehovot
  - Ichilov medical center Tel Aviv, Tel Aviv

IPD SHARING:
Plan to Share IPD: No